CLINICAL TRIAL: NCT06306196
Title: A Phase 2b, Open-label Study to Evaluate the Immunogenicity and Safety of Hecolin® in HIV Positive/Negative Adult Participants Followed by a Randomized, Placebo-controlled, Observer-blind Study to Evaluate the Immunogenicity and Safety of Hecolin® in Children
Brief Title: Immunogenicity and Safety of Hecolin® in HIV Positive/Negative Adults and in Children
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: International Vaccine Institute (Other)
Collaborators: Xiamen Innovax Biotech Co., Ltd (Industry); Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: IVI Hecolin S001
Record Dates: First submitted 2024-02-18; First posted 2024-03-12 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Hepatitis E Virus Infection
MeSH Terms: conditions — Hepatitis E | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Adult participants will receive open-label IP and the PI, study staff and participants will not be blinded to Hecolin® administration.
  For children cohorts, the PI, study staff, and child participants will be blinded as to receipt of the study vaccine or placebo. The unblinded pharmacist preparing the IP as well as the unblinded vaccinator will not be involved in the safety assessment of participants and will be instructed not to comment on the experimental agent to study staff.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (17):
- Group A1 (Three doses of Hecolin®; HIV negative adults aged 18-45 years) (Experimental): Three doses of Hecolin® Recombinant Hepatitis E Vaccine administered at 0, 1 and 6 months to HIV negative participants, age 18-45 years old, 232 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group A2 (Three doses of Hecolin®; HIV positive adults aged 18-45 years) (Experimental): Three doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, 1 and 6 months, to HIV positive participants, age 18-45 years old, 178 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group B1 (Three doses of Hecolin®; healthy adolescents aged 12-17 years) (Experimental): Three doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, 1 and 6 months, to age 12-17 years old, 70 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group B2 (Two doses of Hecolin®; healthy adolescents aged 12-17 years) (Experimental): Two doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, 1 and 6 months) and one dose of Placebo, administered at 1-month timepoint, to age 12-17 years old, 70 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine; Biological: Isotonic Sodium Chloride injection
- Group B3 (Placebo; healthy adolescents aged 12-17 years) (Placebo Comparator): Three doses of Placebo, administered at 0, 1 and 6 months, to age 12-17 years old, 35 participants
  Interventions: Biological: Isotonic Sodium Chloride injection
- Group C1 (Three doses of Hecolin®; healthy children aged 6-11 years) (Experimental): Three doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, 1 and 6 months, to age 6-11 years old, 70 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group C2 (Two doses of Hecolin®; healthy children aged 6-11 years) (Experimental): Two doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0 and 6 months and one dose of Placebo, administered at 1-month timepoint, to age 6-11 years old, 70 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine; Biological: Isotonic Sodium Chloride injection
- Group C3 (Placebo; healthy children aged 6-11 years) (Placebo Comparator): Three doses of Placebo, administered at 0, 1 and 6 months, to age 6-11 years old, 35 participants
  Interventions: Biological: Isotonic Sodium Chloride injection
- Group D1 (Three doses of Hecolin®; healthy children aged 2-5 years) (Experimental): Three doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, 1 and 6 months, to age 2-5 years old, 40 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group D2 (Two doses of Hecolin®; healthy children aged 2-5 years) (Experimental): Two doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0 and 6 months and of Placebo, administered at 1-month timepoint, to age 2-5 years old, 40 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine; Biological: Isotonic Sodium Chloride injection
- Group D3 (Placebo; healthy children aged 2-5 years) (Placebo Comparator): Three doses of Placebo, administered at 0, 1 and 6 months, to age 2-5 years old, 40 participants
  Interventions: Biological: Isotonic Sodium Chloride injection
- Group B4 (Two doses of Hecolin®; healthy children aged 12-17 years) (Experimental): Two doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, and 1 month, to age 12-17 years old, 50 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group B5 (Placebo; healthy children aged 12-17 years) (Experimental): Two doses of Placebo, administered at 0, and 1 month, to age 12-17 years old, 10 participants
  Interventions: Biological: Isotonic Sodium Chloride injection
- Group C4 (Two doses of Hecolin®; healthy children aged 6-11 years) (Experimental): Two doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, and 1 month, to age 6-11 years old, 50 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group C5 (Placebo; healthy children aged 6-11 years) (Experimental): Two doses of Placebo, administered at 0, and 1 month, to age 6-11 years old, 10 participants
  Interventions: Biological: Isotonic Sodium Chloride injection
- Group D4 (Two doses of Hecolin®; healthy children aged 2-5 years) (Experimental): Two doses of Hecolin® Recombinant Hepatitis E Vaccine, administered at 0, and 1 month, to age 2-5 years old, 50 participants
  Interventions: Biological: Hecolin® Recombinant Hepatitis E Vaccine
- Group D5 (Placebo; healthy children aged 2-5 years) (Experimental): Two doses of Placebo, administered at 0, and 1 month, to age 2-5 years old, 10 participants
  Interventions: Biological: Isotonic Sodium Chloride injection

INTERVENTIONS:
Biological: Hecolin® Recombinant Hepatitis E Vaccine — 30㎍/dose, 0.5mL administered intramuscularly
  Arms: Group A1 (Three doses of Hecolin®; HIV negative adults aged 18-45 years); Group A2 (Three doses of Hecolin®; HIV positive adults aged 18-45 years); Group B1 (Three doses of Hecolin®; healthy adolescents aged 12-17 years); Group B2 (Two doses of Hecolin®; healthy adolescents aged 12-17 years); Group B4 (Two doses of Hecolin®; healthy children aged 12-17 years); Group C1 (Three doses of Hecolin®; healthy children aged 6-11 years); Group C2 (Two doses of Hecolin®; healthy children aged 6-11 years); Group C4 (Two doses of Hecolin®; healthy children aged 6-11 years); Group D1 (Three doses of Hecolin®; healthy children aged 2-5 years); Group D2 (Two doses of Hecolin®; healthy children aged 2-5 years); Group D4 (Two doses of Hecolin®; healthy children aged 2-5 years)
Biological: Isotonic Sodium Chloride injection — 0.5mL administered intramuscularly
  Arms: Group B2 (Two doses of Hecolin®; healthy adolescents aged 12-17 years); Group B3 (Placebo; healthy adolescents aged 12-17 years); Group B5 (Placebo; healthy children aged 12-17 years); Group C2 (Two doses of Hecolin®; healthy children aged 6-11 years); Group C3 (Placebo; healthy children aged 6-11 years); Group C5 (Placebo; healthy children aged 6-11 years); Group D2 (Two doses of Hecolin®; healthy children aged 2-5 years); Group D3 (Placebo; healthy children aged 2-5 years); Group D5 (Placebo; healthy children aged 2-5 years)

SUMMARY:
The primary goal of this clinical trial is to demonstrate non-inferiority of 30 µg of Hecolin® in healthy children, compared to healthy adults as measured by seroresponse rates (SR) of anti-HEV IgG titers, 4 weeks after 3 doses (0, 1 and 6 months) and to assess and descriptively compare safety profile data intra and inter age Strata. As secondary objectives, Geometric Mean Concentration (GMC) of anti-HEV IgG ELISA will be evaluated 4 weeks after 3 doses (0, 1 and 6 months) and 4 weeks after 2 doses (0- and 6-months dose) in healthy children. SR and GMC will also be evaluated 24 weeks after 3 doses and 2 doses. The immune response will be compared among adult participants between HIV positive and HIV negative individuals and between virally suppressed and virally unsuppressed HIV positive individuals

DETAILED DESCRIPTION:
The primary objective of the study is to demonstrate immune non-inferiority of 30 µg Hecolin® when given to healthy children (2-17 years) as compared to healthy adults (18-45 years) as measured by seroresponse rates (SR) of anti- HEV IgG ELISA antibody titers, 4 weeks after the 3 doses given at 0, 1- & 6-months. Co-primary objective is to assess safety in each age cohort and descriptively compare lower age cohorts with higher age cohorts. Other immune parameters would be assessed as secondary objectives. Healthy children and adolescents collectively (2-17 years) will be compared for immune non-inferiority with healthy adults (18-45 years) as measured by geometric mean concentration (GMC) of anti-HEV IgG ELISA antibody titers, 4 weeks after the 3 doses given at 0, 1- & 6-months. Among children (2-17 years) 3 doses of Hecolin® given at 0, 1 and 6 months will be compared with 2 doses of Hecolin® given at 1 and 6 months in terms of immune non-inferiority of SR and GMC of anti-HEV IgG ELISA antibody titers. The immune response will be compared between HIV positive and HIV negative adults in terms of SR and GMC as measured by anti-HEV IgG ELISA antibody titers at 4 weeks after completing 3 doses of Hecolin® (0, 1 and 6 months).

A total of 860 participants will be enrolled in the main study and will be divided into 4 age strata; 18-45 years (Cohort A), 12-17 years (Cohort B), 6-11 years (Cohort C) and 2-5 years (Cohort D) having 410, 175, 175 and 100 participants respectively. Cohort A will be further divided into Arm A1 and A2 having 232 HIV -ve and 178 HIV +ve participants respectively. All participants in cohort A will receive intramuscular injection of 3 doses of 30 µg Hecolin® at 0, 1 and 6 months. Cohort B will be further divided into Arm B1, B2 and B3 having 70, 70 and 35 participants respectively. Arm B1 will receive intramuscular injection of 3 doses of 30 µg Hecolin® at 0, 1 and 6 months. Arm B2 will receive intramuscular injection of 2 doses of 30 µg Hecolin® at 0 and 6 months while Arm B3 will receive intramuscular injection of comparator (placebo) intramuscularly at 0, 1 and 6 months. Similarly, Cohort C will be further divided into Arm C1, C2 and C3 having 70, 70 and 35 participants respectively. Arm C1 will receive intramuscular injection of 3 doses of 30 µg Hecolin® at 0, 1 and 6 months. Arm C2 will receive intramuscular injection of 2 doses of 30 µg Hecolin® at 0 and 6 months while Arm C3 will receive intramuscular injection of comparator (placebo) intramuscularly at 0, 1 and 6 months. Cohort D will be further divided into Arm D1, D2 and D3 having 40, 40 and 20 participants respectively. Arm D1 will receive intramuscular injection of 3 doses of 30 µg Hecolin® at 0, 1 and 6 months. Arm D2 will receive intramuscular injection of 2 doses of 30 µg Hecolin® at 0 and 6 months while Arm D3 will receive intramuscular injection of comparator (placebo) intramuscularly at 0,1 and 6 months.

In the main study a total of 6 blood samples for immunogenicity will be collected from all participants at Day 0 (baseline), one month after first vaccination, one month after second vaccination, 6 months after first vaccination, one month after third vaccination, and at 6 months after third vaccination.

Blood samples will be collected at screening and one month after third vaccination from the HIV + arm to document CD4 T cells and HIV Viral load.

Out of the 860 participants enrolled in the main study, 2 additional blood samples after reconsent for the 2-year long term follow up period will be collected at V8 (12 months after 3rd dose) and V9 (24 months after 3rd dose) from any 100 HIV negative adults in Cohort A and from participants in Hecolin arms in Cohorts B, C and D (B1, B2, C1, C2, D1, and D2) for immunogenicity assessment. In the additional 0-1-month dose schedule component/arm, a total of 4 blood samples will be collected from all participants at V2 (Day 0), V3 (28 days after 1st dose), V4 (28 days after 2nd dose), V5 (6 months after 2nd dose), and 2 additional samples will be collected from participants in Hecolin arms in Cohorts B, C and D (B4, C4, and D4) at V6 (12months after 2nd dose), and V7 (24 months after 2nd dose) for immunogenicity assessment.

All participants will be observed at the study site for 30 minutes after each Investigational Product (IP) injection for any reactogenicity events. Local and systemic solicited adverse events will be recorded in a diary card during 7 days after each IP dose while unsolicited adverse events will be recorded during the 4 weeks after each IP injection. Serious adverse events (SAEs), Medically attended adverse events (MAAEs) and Adverse of special interest (AESI) will be recorded during the entire study period i.e., until 6 months post last dose.

ELIGIBILITY:
Inclusion Criteria (healthy participants only):

1. Healthy participants 2 to 45 years of age at enrollment,
2. Participants/Parent(s)/LAR who have voluntarily given informed consent/assent,
3. Participants/Parent(s)/LAR willing to follow the study procedures and available for the entire duration of the study and agrees to the collection of all biospecimens,
4. HIV negative,
5. Not pregnant,
6. Agreement to practice effective contraception for female participants of childbearing potential and non-sterile males until at least 8 months after the first vaccination.
7. Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the first dose of vaccine, and
8. Female participant not currently breastfeeding.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Has received any hepatitis E vaccine in the past,
2. Febrile illness (body temperature ≥ 38°C) or acute illness within 3 days prior to the study vaccination,
3. Known history or allergy to study vaccine components and/or excipients or other medications, or any other allergies or medical history deemed by the investigator to increase the risk of an adverse event if they were to participate in the trial (e.g., Guillain-Barre Syndrome),
4. Major congenital abnormalities which in the opinion of the investigator may affect the participant's participation in the study,
5. Known history of immune function disorders including immunodeficiency diseases (known HIV infection or other immune function disorders) and lupus,
6. Chronic use of systemic steroids (>2 mg/kg/day or >20 mg/day prednisone equivalent for periods exceeding 10 days), cytotoxic or other immunosuppressive drugs within the past 6 weeks,
7. Any abnormality or chronic disease which in the opinion of the investigator might be detrimental to the safety of the participant and interfere with the assessment of the study objectives,
8. Behavioral or cognitive impairment, chronic substance abuse, or psychiatric disease or neural disorders, that, in the opinion of the investigator, could interfere with the participant's ability to participate in the trial,
9. History of splenectomy,
10. History of thrombocytopenia and/or thrombosis, myocarditis or pericarditis or any other significant cardiac condition,
11. With a known bleeding diathesis or any condition that may be associated with a prolonged bleeding time resulting in contraindication for IM injections/blood extractions.,
12. Receipt of blood or blood-derived products in the past 3 months,
13. Receipt of other vaccines from 4 weeks prior to test vaccination or planned to receive any vaccine within 4 weeks of last dose of study vaccine,
14. Concomitantly enrolled or scheduled to be enrolled in another trial,
15. Research staff involved with the clinical study or family/household members of research staff,
16. Body mass index (BMI) of ≥ 40 in adults and for children a BMI- index-for-age is ≥95th percentile, at the time of the screening visit, or
17. As per the Investigator's medical judgement, an individual could be excluded from the study despite meeting all inclusion/exclusion criteria mentioned above.

Inclusion criteria for HIV-positive arm:

1. Adults 18-45 years living with HIV on anti-retroviral (ARV) treatment and willing to have CD4 and viral load measured as per protocol,
2. Able to provide a voluntary signed informed consent,
3. Participants willing to follow the study procedures of the study and available for the entire duration of the study and agrees to the collection of all biospecimens,
4. Agreement to practice effective contraception for female participants of childbearing potential and non-sterile males until at least 3 months after the last vaccination.
5. Has practiced adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to the last dose of vaccine, and
6. Female participant is currently not breastfeeding.

Exclusion Criteria for HIV-positive arm:

An individual who meets any of the following criteria will be excluded from participation in this study:

1. Has received any hepatitis E vaccine in the past,
2. Newly diagnosed HIV-positive (diagnosed on screening) on ARVs for 0-4 weeks (Note: These participants can be re-screened and enrolled once they have been on ARVs for 4 weeks),
3. Febrile illness (body temperature ≥ 38°C) or acute illness within 3 days prior to the study vaccination,
4. Serious adverse reaction to any vaccine, or any component of the investigational vaccine, including a history of anaphylaxis and symptoms of a severe allergic reaction and history of allergies in the past,
5. Current hospitalization,
6. History of inherited blood disorders, heparin-induced thrombocytopenia, or thromboembolic disorders,
7. History of any blood product transfusion up to 6 months before enrolment,
8. Receipt of other vaccines from 4 weeks prior to test vaccination or planned to receive any vaccine within 4 weeks of last dose of study vaccine
9. Currently taking anti-coagulation therapy, or chronic aspirin in the past 3 months,
10. Pregnant or breastfeeding women throughout the study period,
11. Extreme obesity (defined as BMI of 40 kg/m2 or higher),
12. Chronic kidney disease requiring dialysis,
13. Liver disease (Note mild chronic liver disease is not an exclusion criterion),
14. Participants with acquired or hereditary immunodeficiencies other than HIV,
15. History of hereditary, idiopathic, or acquired angioedema,
16. No spleen or functional asplenia,
17. Platelet disorder or other bleeding disorder that may cause injection contraindication,
18. Chronic use (more than 14 continuous days) of any medications that may be associated with impaired immune responsiveness including, but not limited to, systemic corticosteroids exceeding 10 mg/day of prednisone equivalent, allergy injections, immunoglobulin, interferon, or immunomodulators. The use of low dose topical, ophthalmic, inhaled, and intranasal steroid preparations will be permitted,
19. According to the judgement of the investigator, the participant has any other factors that might interfere with the results of the clinical trial or pose additional risk due to participation in the study,
20. Assessed by the Investigator to be unable or unwilling to comply with the requirements of the protocol

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1040 (Estimated)
Dates: Start 2024-04-04 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Seroresponse rate | 4 weeks post third dose of Hecolin®
  Seroresponse rate (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post third dose of Hecolin® administered at 0, 1 and 6 months to healthy children (2-17 years) as compared to healthy adults (18-45 years)
Proportion of immediate adverse events | Within 30 minutes post each dose of vaccination
  Proportion of immediate adverse events within 30 minutes post each dose of vaccination in all study participants
Proportion of solicited local and systemic adverse events | Within 7 days post each dose
  Proportion of solicited local and systemic adverse events within 7 days post each dose of vaccination in all study participants
Proportion of unsolicited adverse events | Within 28 days post each dose
  Proportion of unsolicited adverse events within 28 days post each dose of vaccination in all study participants
Proportion of SAEs, MAAEs and AESIs | Post dose 1 until 6 months post last dose
  Proportion of Serious adverse events (SAEs), Medically attended adverse events (MAAEs) and Adverse events of special interest (AESIs) post dose 1 until 6 months post last dose of vaccination

SECONDARY OUTCOMES:
GMC of anti-HEV IgG | 4 weeks post third dose
  GMC of anti-HEV IgG at 4 weeks post third dose of Hecolin® administered at 0, 1 and 6 months to healthy children (2-17 years) as compared to healthy adults (18-45 years)
SR | 4 weeks post two doses of Hecolin®
  SR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) 4 weeks post two doses of Hecolin® administered at 0, and 6 months as compared to three doses of Hecolin® administered at 0, 1 and 6 months to healthy children (2-17 years)
GMC of anti-HEV IgG | 4 weeks post two doses of Hecolin®
  GMC of anti-HEV IgG at 4 weeks post two doses of Hecolin® administered at 0, and 6 months as compared to three doses of Hecolin® administered at 0, 1 and 6 months to healthy children (2-17 years)
SR and GMC of anti-HEV IgG | 4 weeks post third dose of Hecolin®
  SR and GMC of anti-HEV IgG at 4 weeks post third dose of Hecolin® administered at 0, 1 and 6 months in healthy older children (6-17 years) and healthy adults (18-45 years)
SR | 24 weeks post two doses of Hecolin®
  SR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 24 weeks post two doses of Hecolin® administered at 0, and 6 months as compared to three doses of Hecolin® administered at 0, 1 and 6 months to healthy child
GMC of anti-HEV IgG | 24 weeks post two doses of Hecolin®
  GMC of anti-HEV IgG at 24 weeks post two doses of Hecolin® administered at 0, and 6 months as compared to three doses of Hecolin® administered at 0, 1 and 6 months to healthy children (2-17 years)
SR | 4 weeks post third dose of Hecolin®
  SR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post third dose of Hecolin® administered at 0, 1 and 6 months to HIV-positive adults as compared to HIV-negative healthy adults (18-45 years)
GMC of anti-HEV IgG | 4 weeks post third dose of Hecolin®
  GMC of anti-HEV IgG at 4 weeks post third dose of Hecolin® administered at 0, 1 and 6 months to HIV-positive adults as compared to HIV-negative healthy adults (18-45 years)
SR | 4 weeks post third dose of Hecolin®
  SR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post third dose of Hecolin® administered at 0, 1 and 6 months to virally suppressed (CD4 count < 350) and virally unsuppressed (CD4 count ≥ 350) HIV-positive adults (18-45 years)
GMC of anti-HEV IgG | 4 weeks post third dose of Hecolin®
  MC of anti-HEV IgG at 4 weeks post third dose of Hecolin® administered at 0, 1 and 6 months to virally suppressed (CD4 count < 350) and virally unsuppressed (CD4 count ≥ 350) HIV-positive adults (18-45 years)
SR | 4 weeks post first, second and third dose of Hecolin® /Placebo
  SR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 4 weeks post first, second and third dose of Hecolin® /Placebo administered at 0, 1 and 6 months in healthy children (12-17 years), (6-11 years), (2-5 years) and adults (18-45 years) individually
GMC of anti-HEV IgG | 4 weeks post first, second and third dose of Hecolin® /Placebo
  GMC of anti-HEV IgG at 4 weeks post first, second and third dose of Hecolin® /Placebo administered at 0, 1 and 6 months in healthy children (12-17 years), (6-11 years), (2-5 years) and adults (18-45 years) individually
SR and GMC of anti-HEV IgG | 4 weeks post first, second and third dose of Hecolin® /Placebo
  SR and GMC of anti-HEV IgG at 4 weeks post first, second and third dose of Hecolin® /Placebo administered at 0, 1 and 6 months in healthy children (12-17 years), (6-11 years), (2-5 years) and adults (18-45 years) collectively and individually as per sero- status at baseline.
GMC of anti-HEV IgG for additional 0-1 dose schedule | 4 weeks post first, second of Hecolin
  GMC of anti-HEV IgG at 4 weeks post two doses of Hecolin® administered at 0 and 1 months as compared to three doses of Hecolin® administered at 0, 1 and 6 months to healthy children (2-17 years)
GMC of anti-HEV IgG for additional 0-1 dose schedule | 4 weeks post first, second and third dose of Hecolin® /Placebo
  SR and GMC of anti-HEV IgG in paired sera at 4 weeks post each dose of Hecolin® /Placebo when administered two doses at 0 and 1 months or at 0 and 6 months or three doses at 0, 1 and 6 months in individual age groups in healthy children (12 - 17 years, 6 - 11 years, and 2 - 5 years) or three doses at 0, 1 and 6 months in adults (18 - 45 years).
SR and GMC of anti-HEV IgG for additional 0-1 dose schedule | 4 weeks post first, second and third dose of Hecolin® /Placebo
  SR and GMC of anti-HEV IgG in paired sera at 4 weeks post each dose of Hecolin® /Placebo when administered two doses at 0 and 1 months or at 0 and 6 months or three doses at 0, 1 and 6 months in individual age groups in healthy children (12 - 17 years, 6 - 11 years, and 2 - 5 years) or three doses at 0, 1 and 6 months in adults (18 - 45 years).
SR and GMC of anti-HEV IgG for additional 0-1 dose schedule | 24 weeks post two doses of Hecolin®
  SR (antibody response greater than four times or more increase of anti-HEV IgG in paired sera) at 24 weeks post two doses of Hecolin® administered at 0-, and 1- month in healthy children (2-17 years).
SR and GMC of anti-HEV IgG for additional long-term follow up component | 1 and 2 years post two doses of Hecolin®
  SR and GMC (defined as the percentage of participants with anti-HEV IgG antibodies above the detection limit, assessed at 1 year and 2 years post two doses of Hecolin® administered in healthy children (2-17 years) at 0- & 6-months or at 0- & 1-month or post 3 doses (0, 1 & 6 month) in healthy children (2-17 years) and healthy adults (18-45 years)

OTHER OUTCOMES:
SR and GMC of anti-HEV IgG | 4 weeks post first, second and third dose of Hecolin® /Placebo
  SR and GMC of anti-HEV IgG at 4 weeks post first, second and third dose of Hecolin® /Placebo administered at 0, 1 and 6 months in healthy children (12-17 years), (6-11 years), (2-5 years) and adults (18-45 years) collectively and individually as per gender distribution
Safety in all participants as per gender distribution and serostatus | 1. Within 30 minutes post each dose of vaccination. 2. Within 7 days post each dose of vaccination. 3. Within 28 days post each dose of vaccination. 4.Until 6 months post last dose of vaccination.
  1. Proportion of immediate adverse events within 30 minutes post each dose of vaccination in all study participants.
  2. Proportion of solicited local and systemic adverse events within 7 days post each dose of vaccination in all study participants.
  3. Proportion of unsolicited adverse events within 28 days post each dose of vaccination in all study participants.
  4. Proportion of Serious adverse events (SAEs), Medically attended adverse events (MAAEs) and Adverse of special interest (AESI) until 6 months post last dose of vaccination.
Safety profile intra and inter age strata | 1. Within 30 minutes post each dose of vaccination. 2. Within 7 days post each dose of vaccination. 3. Within 28 days post each dose of vaccination. 4.Until 6 months post last dose of vaccination
  1. Proportion of immediate adverse events within 30 minutes post each dose of vaccination in all study participants.
  2. Proportion of solicited local and systemic adverse events within 7 days post each dose of vaccination in all study participants.
  3. Proportion of unsolicited adverse events within 28 days post each dose of vaccination in all study participants.
  4. Proportion of Serious adverse events (SAEs), Medically attended adverse events (MAAEs) and Adverse events of special interest (AESI) post dose 1 until 6 months post last dose of vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Tarun Saluja, Principal Investigator — International Vaccine Institute; Sanet Aspinall, Principal Investigator — Ardent Consulting (Pty) Ltd; Elizabeth Hellström, Principal Investigator — Be Part Research; Maphoshane Nchabeleng, Principal Investigator — MeCRU Clinical Research Unit; Essack Mitha, Principal Investigator — Newtown Clinical Research Centre
Locations (3):
- South Africa (3):
  - MeCRU Clinical Research Unit, Ga-Rankuwa
  - Newtown Clinical Research Centre, Johannesburg
  - Be Part Research, Paarl

IPD SHARING:
Plan to Share IPD: No